CLINICAL TRIAL: NCT01258933
Title: Ofatumumab for Residual Disease and Maintenance Following Chemotherapy or Chemoimmunotherapy in Patients With Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL)
Brief Title: Ofatumumab for Minimal Residual Disease (MRD) and Maintenance Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0266; NCI-2011-00274 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-12-09; First posted 2010-12-13 (Estimated); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Leukemia; Lymphoma
Keywords: Leukemia; Chronic Lymphocytic Leukemia; CLL; Lymphoma; Small Lymphocytic Lymphoma; SLL; Ofatumumab
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ofatumumab (Experimental): Ofatumumab 300 mg dose 1, then 1,000 mg weekly * 7, (treatment) then 1,000 mg every 2 months beginning on week 12 for a total of 2 years of treatment or until progression (maintenance) of disease. The follow-up period will be the period after completion of maintenance.
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — 300 mg Dose 1, then 1,000 mg weekly x 7, (treatment) then 1,000 mg every 2 months beginning on week 12
  Other Names: Arzerra

SUMMARY:
The goal of this clinical research study is to find out if ofatumumab can control CLL or SLL that is left after chemotherapy or chemoimmunotherapy. The safety of the drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Ofatumumab is designed to bind to the surface of some white blood cells (B-cells) and to kill these cells. It can destroy cancer cells that come from B-cells, and can be used to treat cancers of B-cells such as B-CLL.

Study Drug Administration If you are found to be eligible to take part in this study, you will receive ofatumumab up to 20 times during this study. You will receive 8 weekly infusions and then an infusion every 2 months for 2 years or until the disease gets worse. You will receive ofatumumab by vein over about 6 ½ hours the first time and over 4 hours for all the following infusions. The first infusion will be the smallest dose. The second and later infusions will be 3 times larger than the first.

Before you receive the study drug each time, you will receive Tylenol (acetaminophen) by mouth to reduce the risk of fever. You will receive Benadryl (diphenhydramine) by mouth or vein and prednisolone (a steroid) by vein over about 30 minutes to reduce the risk of an allergic reaction or an infusion reaction.

During the infusions, you will be monitored closely. You will be expected to stay in clinic for about 71/2 hours on the day of the first infusion and 5 hours for all other infusions.

You will be seen at MD Anderson for mandatory visits for enrollment, ofatumumab infusions, for response assessment after 8 weekly ofatumumab doses (Month 3), during maintenance every 6 months and for follow-up at least once a year. Your local doctor may perform other visits and laboratory studies.

If you decide to have your local doctor perform study visits and laboratory studies, a letter will be sent to your doctor, describing your participation in this study and asking for your doctor's agreement to help manage your care.

Study Visits

The following tests and procedures will be performed every other week during Weeks 1- 8 (Weeks 1, 3, 5 and 7):

You will have a complete physical exam including measurement of your vital signs.

Your medical history will be recorded. Blood (about 2 teaspoons) will be drawn for routine tests.

Starting at Month 3, you will have the following tests and procedures every 2 Months:

You will have a complete physical exam including measurement of your vital signs.

Your medical history will be recorded. Blood (about 2 teaspoons) will be drawn for routine tests.

Starting at Month 3, you will also have the following tests and procedures every 6 months, in addition to the ones performed every 2 months:

Blood (about an additional 1 teaspoon) will be drawn for other routine tests. You may have CT scans to check the status of the disease, if your doctor thinks that this test is needed (at Month 3 only).

You will have a bone marrow aspirate/biopsy to check the status of the disease.

Additional Information Depending on the results of your hepatitis tests performed at the screening visit, you may have additional hepatitis tests. The study staff will tell you if you will have these tests performed. If you do have the additional hepatitis tests, blood (about 2 teaspoons) will be drawn during Months 3-24. The blood will be drawn at the same time of the routine blood draws to prevent unnecessary needle sticks.

Length of Study You may continue taking the study drug for up to 20 doses (up to 24 months). You will no longer be able to take the study drug if the disease gets worse or intolerable side effects occur.

Your participation on the study will be over once you have completed the follow-up visits, which will last until you begin receiving any other treatment.

Follow Up Visits Every 3 Months You will have a complete physical exam including measurement of your vital signs.

Your medical history will be recorded. Blood (about 2 teaspoons every 3 months, about 1 teaspoon every 6 months) will be drawn for routine tests.

If your doctor thinks it is needed, blood (about 2 teaspoons) will be drawn for hepatitis testing.

Every 6 Months, you will have a bone marrow aspirate/biopsy to check the status of the disease.

This is an investigational study. Ofatumumab is FDA approved for CLL resistant to standard chemotherapy. Ofatumumab's use in patients with residual CLL or SLL is investigational.

Ofatumumab will be provided at no cost to you while you are on the study.

Up to 42 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CD20+ chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) treated with chemotherapy or chemoimmunotherapy: Post-frontline therapy, patients must have non-progressing disease and be 4 months to 1 year post treatment. Post-treatment for relapsed CLL, eligible patients must have non-progressing disease and be 3 months to 1 year post treatment.
2. Patients (CR, nPR, or PR at enrollment) must have measurable disease, which may include MRD by 4-color flow cytometry.
3. Adequate renal and hepatic function (creatinine < 2 mg/dL, bilirubin < 2 mg/dL). Patients with renal or liver dysfunction due to organ infiltration by lymphocytes may be eligible after discussion with the study chairman. Patients with Gilbert's syndrome are eligible.
4. Age >/= 18 years.
5. ECOG performance status of 0-2.
6. Provide informed consent indicating patient is aware of the investigational nature of this study according to the policies of the MDACC IRB.
7. Patients of childbearing potential (females who have not been postmenopausal for at least 12 consecutive months or who have not undergone previous surgical sterilization or males who have not been surgically sterilized) must be willing to practice birth control during the study.

Exclusion Criteria:

1. Positive serology for Hepatitis B virus (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HB DNA test will be performed and if positive the subject will be excluded.
2. Concurrent chemotherapy, radiotherapy, or immunotherapy, including other monoclonal antibodies. Localized radiotherapy to an area not comprising bone marrow function does not apply.
3. Active infection or significant medical illness, including current active hepatic or biliary disease (with exception of patients with asymptomatic gallstones, liver involved with CLL or stable chronic liver disease per investigator assessment).
4. Pregnant and breastfeeding females are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-07-06 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G Wierda, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ofatumumab
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ofatumumab
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 70 [64 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Objective Response
Description: Response assessment according to 2008 International Working Group for CLL (IWCLL), prior to 9th dose of ofatumumab (prior to first bimonthly dose). Responses of (complete remission (CR) conversion to minimal residual disease (MRD) negative, partial remission (PR) conversion to nodular partial remission nPR or CR, and nPR conversion to complete remission (CR)) evaluated by physical examination, CBC, CT of chest, abdomen, pelvis, and bone marrow aspirate and biopsy with evaluation of residual disease (MRD) by 4-color flow cytometry.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 4
Participants | 0

2. Secondary Outcome: Time-to-Treatment Failure (TTF)
Description: Time from date of treatment start until the date of failure or death from any cause.
Time Frame: Start of study drug up to approximately 1 year and 7 months.
Measure: Median (Full Range); unit: Months
Arm/Group | Ofatumumab
Number analyzed (Participants) | 4
Months | 8.6 [1.6 to 12.7]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Time from date of treatment start until the date of progression or death from leukemia.
Time Frame: Start of study drug up to approximately 7 years and 6 months.
Measure: Median (Full Range); unit: Months
Arm/Group | Ofatumumab
Number analyzed (Participants) | 4
Months | 26.0 [25.1 to 90.0]

ADVERSE EVENTS:
Time Frame: Adverse Events monitored monthly until follow-up, assessed up to 3 years. Mortality was monitored up to approximately 13 years, 3 months.
Arm/Group | Ofatumumab
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ofatumumab (N=4)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Splenectomy (Surgical and medical procedures) | 1 (1)
Infusion reaction (General disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
edema (General disorders) | 2 (2)
fatigue (General disorders) | 2 (2)
fever (General disorders) | 3 (3)
Flu-like Syndrome (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2011-12-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT01258933/Prot_SAP_001.pdf
  • Informed Consent Form (2011-07-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT01258933/ICF_000.pdf